CLINICAL TRIAL: NCT07400341
Title: A Randomized Phase II Study of Romiplostim vs. rhTPO for Platelet Engraftment After Allo-HSCT in Patients With MDS and Aplastic Anemia (PROMPT)
Brief Title: Romiplostim Versus rhTPO for Platelet Engraftment After Transplant in MDS and AA
Acronym: PROMPT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOOCHOW-WXJ-2025-1294
Record Dates: First submitted 2026-01-19; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: MDS (Myelodysplastic Syndrome); Aplastic Anemia (AA)
Keywords: Romiplostim; Recombinant Human Thrombopoietin (rhTPO); Platelet Engraftment; Delayed Platelet Recovery
MeSH Terms: conditions — Anemia, Refractory, with Excess of Blasts; Anemia, Aplastic | interventions — romiplostim; Thrombopoietin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- rhTPO (Recombinant Human Thrombopoietin) (Active Comparator): Participants will receive subcutaneous rhTPO injections at a fixed dose of 15000 U once daily, beginning on transplant day +4. Treatment continues until the platelet count is ≥50×10⁹/L without transfusion for 7 days, until day +60 post-transplant, or for a maximum of 8 weeks, whichever occurs first.
  Interventions: Drug: Recombinant Human Thrombopoietin
- Romiplostim (Experimental): Participants will receive subcutaneous Romiplostim injections at a starting dose of 5.0 µg/kg once weekly, beginning on transplant day +4. The dose will be adjusted weekly based on platelet counts. Treatment continues until the platelet count is ≥50×10⁹/L without transfusion for 7 days, until day +60 post-transplant, or for a maximum of 8 weeks, whichever occurs first.
  Interventions: Drug: Romiplostim

INTERVENTIONS:
Drug: Romiplostim — Romiplostim is a thrombopoietin receptor agonist (TPO-RA) that stimulates platelet production. It is a fusion protein (peptibody) that binds to and activates the TPO receptor, promoting megakaryocyte proliferation and differentiation. In this study, it is administered as a subcutaneous injection once weekly.
  Other Names: TPO-RA
  Arms: Romiplostim
Drug: Recombinant Human Thrombopoietin — Recombinant human thrombopoietin is a cytokine that stimulates platelet production by binding to the TPO receptor on megakaryocytes. In this study, it is administered as a subcutaneous injection once daily.
  Other Names: rhTPO
  Arms: rhTPO (Recombinant Human Thrombopoietin)

SUMMARY:
This study is for adults aged 18-65 with myelodysplastic syndrome (MDS) or severe aplastic anemia (AA) who are scheduled to receive a donor stem cell transplant (allogeneic hematopoietic stem cell transplant). After the transplant, it is critical for the body to start making its own blood cells again. A common and serious problem is a delay in the recovery of platelets (the cells that help stop bleeding), which increases the risk of bleeding, infection, and death.

This study aims to see if a new treatment can help platelets recover faster and more safely after transplant. We are comparing two drugs:

Romiplostim: A long-acting injection given just once a week. rhTPO (Recombinant Human Thrombopoietin): A standard injection given every day. Both drugs are designed to help the body make more platelets. The main question is whether the once-weekly romiplostim works as well or better than the daily rhTPO, and if it is safe.

About 66 patients will participate. By random chance (like flipping a coin), each participant will be assigned to receive either romiplostim or rhTPO. The treatment will start a few days after the transplant and continue until platelets recover to a safe level or for up to 8 weeks. Doctors will closely monitor all participants for 100 days to track platelet recovery, need for transfusions, side effects, and overall health.

DETAILED DESCRIPTION:
This is a prospective, single-center, randomized, open-label, parallel-controlled Phase II clinical trial. The primary objective is to provide a preliminary efficacy estimate and evaluate the safety of romiplostim compared to recombinant human thrombopoietin (rhTPO) for promoting platelet engraftment following allogeneic hematopoietic stem cell transplantation (allo-HSCT) in patients with myelodysplastic syndrome (MDS) or aplastic anemia (AA).

Study Design and Population:

The study will enroll approximately 74 patients to achieve 66 evaluable subjects, randomized in a 1:1 ratio to the romiplostim group or the rhTPO group. Randomization will be stratified by the underlying disease (MDS vs. AA). Eligible patients are aged 18-65 years, diagnosed with MDS or severe/very severe AA (SAA/VSAA), and are candidates for allo-HSCT from a matched sibling, haploidentical, or unrelated donor (including cord blood). Key inclusion criteria require a platelet count <20×10⁹/L with transfusion dependence between day +4 and day +10 post-transplant. Major exclusion criteria include uncontrolled active infection, significant history of thrombosis, active transplant-associated thrombotic microangiopathy (TA-TMA), pre-transplant bone marrow fibrosis ≥ MF-2 grade, and known allergy to the study drugs.

Interventions:

Experimental Group (n≈33): Romiplostim administered subcutaneously at a starting dose of 5.0 µg/kg once weekly, beginning on transplant day +4. Subsequent doses (from day +18) will be adjusted weekly based on platelet counts.

Active Control Group (n≈33): rhTPO administered subcutaneously at a fixed dose of 15000 U once daily, beginning on transplant day +4.

Treatment for both groups continues until the platelet count is ≥50×10⁹/L without transfusion support for 7 consecutive days, until day +60 post-transplant, or for a maximum of 8 weeks, whichever occurs first. All patients will receive standardized transplant supportive care.

Endpoints:

Primary Endpoints:

Platelet engraftment time, defined as the first of three consecutive days with a platelet count ≥20×10⁹/L without platelet transfusion in the preceding 7 days.

Incidence of ≥ Grade 3 adverse events (AEs) within 100 days post-transplant, with specific focus on graft-versus-host disease (GVHD) and thrombotic events.

Secondary Endpoints: Platelet engraftment rate at day 60 (≥50×10⁹/L), total platelet transfusion units from day 0 to 60, overall survival (OS), progression-free survival (PFS), and non-relapse mortality (NRM).

Exploratory Endpoints: Immune reconstitution (lymphocyte subsets), megakaryocyte-related biomarkers, and a pharmacoeconomic evaluation.

Oversight and Safety:

An Independent Data Safety Monitoring Committee (DSMB) will be established to periodically review accumulated safety data. Safety will be actively monitored through weekly clinical and laboratory assessments during the treatment period, with specific focus on thrombotic events, GVHD, and potential clonal evolution. The study will be conducted at the Department of Hematology, The First Affiliated Hospital of Soochow University, China, following approval by its institutional Ethics Committee.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years (inclusive).
2. Diagnosis of Myelodysplastic Syndrome (MDS) per WHO criteria, or Severe/Very Severe Aplastic Anemia (SAA/VSAA) per Camitta criteria, and deemed eligible for allogeneic hematopoietic stem cell transplantation (allo-HSCT).
3. Planned to receive allo-HSCT from a matched sibling, haploidentical, or unrelated donor (including cord blood).
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
5. Persistent platelet count <20×10⁹/L with platelet transfusion dependence between post-transplant days +4 and +10. Transfusion dependence is defined as platelet count not doubling within 24-48 hours after transfusion or ongoing need for prophylactic transfusion.
6. Adequate cardiac, hepatic, and renal function as required for transplantation, per investigator assessment.
7. Voluntary participation with written informed consent obtained prior to any study-specific procedures.

Exclusion Criteria:

1. Active, uncontrolled bacterial, fungal, or viral infection at the time of enrollment.
2. History of arterial thrombosis, or venous thromboembolism within the past 6 months (unless cured or stable for over 6 months).
3. Active transplant-associated thrombotic microangiopathy (TA-TMA).
4. Pre-transplant bone marrow biopsy showing fibrosis grade ≥ MF-2 (according to WHO criteria).
5. Known hypersensitivity to Romiplostim, recombinant human thrombopoietin (rhTPO), or any of their excipients.
6. Pregnant or lactating women.
7. Women of childbearing potential or men with partners of childbearing potential who are unwilling to use highly effective contraception during the study period and for at least 3 months after the last dose of study drug.
8. Any other condition that, in the opinion of the investigator, would make the patient unsuitable for participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of Platelet Engraftment by Day +60 (Platelets ≥50×10^9/L without transfusion for 7 consecutive days) | From the start of transplantation until Day 60 post-transplant (or until the engraftment criterion is met).
  To preliminarily evaluate and compare the efficacy of romiplostim versus rhTPO in promoting platelet recovery after allo-HSCT. Engraftment is defined as achieving a platelet count ≥50×10^9/L without transfusion support for 7 consecutive days.
Incidence of ≥ Grade 3 Adverse Events within 100 Days Post-Transplant (including GVHD and thrombotic events) | From the start of transplantation until Day 100 post-transplant.
  To assess and compare the safety profile between romiplostim and rhTPO, focusing on severe adverse events. Events of special interest include acute/chronic GVHD (graded per NIH criteria) and thrombotic events (e.g., TA-TMA, deep vein thrombosis).

SECONDARY OUTCOMES:
60-Day Platelet Engraftment Rate | At Day 60 post-transplant.
  Proportion of participants achieving platelet engraftment (defined as platelet count ≥50×10⁹/L) by Day 60 post-transplant without platelet transfusion support.
Platelet Transfusion Requirements (Days 0-60) | From Day 0 (day of transplant) to Day 60 post-transplant.
  Total number of platelet transfusion units (including both prophylactic and therapeutic transfusions) administered from Day 0 (day of transplant) to Day 60 post-transplant.
Overall Survival (OS) | From date of transplant until death from any cause, assessed up to 2 years.
  Time from the date of transplant until death from any cause. Participants alive at the end of follow-up will be censored.
Progression-Free Survival (PFS) | From date of transplant until disease progression/relapse or death from any cause, assessed up to 2 years.
  Time from the date of transplant until disease progression/relapse or death from any cause, whichever occurs first.
Non-Relapse Mortality (NRM) | From date of transplant until death from non-relapse causes, assessed up to 2 years.
  Cumulative incidence of death from causes other than disease relapse/progression.

OTHER OUTCOMES:
Immune reconstitution | At post-transplant day +30 and day +100 (±7 days)
  Immune reconstitution (lymphocyte subsets, such as CD4+/CD8+ T cells, NK cells, B cell counts)
Megakaryocyte Count and Maturity in Bone Marrow | At post-transplant day +14 (±3 days) and day +28 (±3 days)
  Assessment of megakaryocyte quantity and maturation stage in bone marrow post-transplant, as measured by flow cytometry for CD41+/CD61+ (total count) and CD41+/CD61+/CD36+ (maturity)
Serum Thrombopoietin (TPO) Level | At post-transplant day +14 (±3 days) and day +28 (±3 days)
  Measurement of serum Thrombopoietin (TPO) concentration post-transplant.
From the start of transplantation (Day 0) until Day +100 post-transplant | From the start of transplantation (Day 0) until Day +100 post-transplant.
  Comparison of total direct medical costs between treatment groups, including costs of inpatient hospitalization and study drug administration (romiplostim or rhTPO). Costs will be calculated in Chinese Yuan (CNY) and reported as mean cost per participant.
Incremental Cost-Effectiveness Ratio (ICER) | From the start of transplantation (Day 0) until Day +100 post-transplant
  The incremental cost per additional unit of health benefit (e.g., per additional patient achieving platelet engraftment by Day 60) will be calculated by comparing the difference in total costs to the difference in the primary efficacy outcome (rate of platelet engraftment) between groups.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Department of Hematology, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
Individual de-identified participant data that underlie the reported results may be shared upon reasonable request after article publication, subject to a data use agreement.

REFERENCES:
- [Background] Scordo M, Gilbert LJ, Hanley DM, Flynn JR, Devlin SM, Nguyen LK, Ruiz JD, Shah GL, Sauter CS, Chung DJ, Landau HJ, Lahoud OB, Lin RJ, Dahi PB, Perales MA, Giralt SA, Soff GA. Open-label pilot study of romiplostim for thrombocytopenia after autologous hematopoietic cell transplantation. Blood Adv. 2023 Apr 25;7(8):1536-1544. doi: 10.1182/bloodadvances.2022007838. PMID 36409612
- [Background] Xie C, Zhao H, Bao X, Fu H, Lou L. Pharmacological characterization of hetrombopag, a novel orally active human thrombopoietin receptor agonist. J Cell Mol Med. 2018 Nov;22(11):5367-5377. doi: 10.1111/jcmm.13809. Epub 2018 Aug 29. PMID 30156363
- [Background] Wang R, Cai J, Chen Z, Tian H, Cong D, Bai Y, Zhang W. Recombinant human thrombopoietin does not promote platelet engraftment in newly diagnosed multiple myeloma patients following autologous stem cell transplantation. Sci Rep. 2025 Feb 13;15(1):5393. doi: 10.1038/s41598-025-89535-7. PMID 39948233
- [Background] Wang H, Huang M, Zhao Y, Qi JQ, Chen C, Tang YQ, Qiu HY, Fu CC, Tang XW, Wu DP, Ruan CG, Han Y. Recombinant Human Thrombopoietin Promotes Platelet Engraftment and Improves Prognosis of Patients with Myelodysplastic Syndromes and Aplastic Anemia after Allogeneic Hematopoietic Stem Cell Transplantation. Biol Blood Marrow Transplant. 2017 Oct;23(10):1678-1684. doi: 10.1016/j.bbmt.2017.06.010. Epub 2017 Jun 19. PMID 28642072
- [Background] Han TT, Xu LP, Liu DH, Liu KY, Wang FR, Wang Y, Yan CH, Chen YH, Sun YQ, Ji Y, Wang JZ, Zhang XH, Huang XJ. Recombinant human thrombopoietin promotes platelet engraftment after haploidentical hematopoietic stem cell transplantation: a prospective randomized controlled trial. Ann Hematol. 2015 Jan;94(1):117-28. doi: 10.1007/s00277-014-2158-1. Epub 2014 Jul 30. PMID 25069650
- [Background] Blumberg N, Heal JM, Phillips GL, Phipps RP. Platelets--to transfuse or not to transfuse. Lancet. 2012 Oct 13;380(9850):1287-9. doi: 10.1016/S0140-6736(12)60983-0. Epub 2012 Aug 8. No abstract available. PMID 22877505
- [Background] Bolwell B, Pohlman B, Sobecks R, Andresen S, Brown S, Rybicki L, Wentling V, Kalaycio M. Prognostic importance of the platelet count 100 days post allogeneic bone marrow transplant. Bone Marrow Transplant. 2004 Feb;33(4):419-23. doi: 10.1038/sj.bmt.1704330. PMID 14688814
- [Background] Kuzmina Z, Eder S, Bohm A, Pernicka E, Vormittag L, Kalhs P, Petkov V, Stary G, Nepp J, Knobler R, Just U, Krenn K, Worel N, Greinix HT. Significantly worse survival of patients with NIH-defined chronic graft-versus-host disease and thrombocytopenia or progressive onset type: results of a prospective study. Leukemia. 2012 Apr;26(4):746-56. doi: 10.1038/leu.2011.257. Epub 2011 Sep 16. PMID 21926960
- [Background] Kanda Y, Chiba S, Hirai H, Sakamaki H, Iseki T, Kodera Y, Karasuno T, Okamoto S, Hirabayashi N, Iwato K, Maruta A, Fujimori Y, Furukawa T, Mineishi S, Matsuo K, Hamajima N, Imamura M. Allogeneic hematopoietic stem cell transplantation from family members other than HLA-identical siblings over the last decade (1991-2000). Blood. 2003 Aug 15;102(4):1541-7. doi: 10.1182/blood-2003-02-0430. Epub 2003 Apr 24. PMID 12714500
- [Background] Yamazaki R, Kuwana M, Mori T, Okazaki Y, Kawakami Y, Ikeda Y, Okamoto S. Prolonged thrombocytopenia after allogeneic hematopoietic stem cell transplantation: associations with impaired platelet production and increased platelet turnover. Bone Marrow Transplant. 2006 Sep;38(5):377-84. doi: 10.1038/sj.bmt.1705444. PMID 16915226
- [Background] Mohty M, Kuentz M, Michallet M, Bourhis JH, Milpied N, Sutton L, Jouet JP, Attal M, Bordigoni P, Cahn JY, Boiron JM, Blaise D; Societe Francaise de Greffe de Moelle et de Therapie Cellulaire (SFGM-TC). Chronic graft-versus-host disease after allogeneic blood stem cell transplantation: long-term results of a randomized study. Blood. 2002 Nov 1;100(9):3128-34. doi: 10.1182/blood.V100.9.3128. PMID 12384409
- [Result] Huang XJ. Current status of haploidentical stem cell transplantation for leukemia. J Hematol Oncol. 2008 Dec 31;1:27. doi: 10.1186/1756-8722-1-27. PMID 19117511

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-12-24): https://cdn.clinicaltrials.gov/large-docs/41/NCT07400341/Prot_SAP_000.pdf